CLINICAL TRIAL: NCT04571125
Title: A Study With Multimodal Neurobiological Approaches to Explore the Interactions Between Monoamine Transporter Genes and Environmental Factors on Attention Deficit Hyperactivity Disorder.
Brief Title: Multimodal Neurobiological Approaches to Explore the Gene-Environment Interactions in ADHD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201912085RINA
Record Dates: First submitted 2020-08-27; First posted 2020-09-30 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2023-06

CONDITIONS: Monoamine Transporter Genes; Environmental Factors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA, plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADHD GROUP: Subjects with clinical diagnosis of ADHD according to the DSM-V criteria
- TD GROUP: Typically development controls without lifetime diagnosis with ADHD

SUMMARY:
Previous studies have demonstrated significant associations of attention-deficit hyperactivity disorder (ADHD) with monoamine transporter genes, including dopamine transporter gene (DAT1), norepinephrine transporter gene (SLC6A2), and serotonin transporter gene (SLC6A4) as well as the important role of environmental factors in the pathogenesis of ADHD. Hence, investigating how genes and environments interact with each other may contribute to the understanding of the pathophysiological mechanisms of ADHD. In this 3-year project, investigators will explore the complex gene-environment interplay in ADHD with multimodal neurobiological approaches, including neuropsychology, neuroimaging, and metabolites, in order to identify the crucial pathophysiological pathways from genes to the brain.

DETAILED DESCRIPTION:
In the present project, investigators aim to explore the complex gene-environment interplay in children with ADHD to identify the crucial pathophysiological pathways from genes to the brain. To achieve our objective, investigators will use multimodal neurobiological approaches to effectively resolve the four major challenges in exploring gene-environment interactions on ADHD.

1. investigators will use multiple levels of neurobiological approaches to identify the interactions between monoamine transporter genes and environment on ADHD, including neuropsychology, neuroimaging, and neuroactive metabolites in plasma, which will provide larger effects than clinical diagnosis.
2. investigators will employ correlation analyses to test for the presence of correlations between the monoamine transporter genotypes and the environmental factors.
3. investigators will use both categorical (diagnosis of ADHD) and dimensional (inattention and hyperactivity-impulsivity symptoms of ADHD) approaches to assess the interaction effects between monoamine transporter genes and environment.
4. investigators will conduct interactions with ageitems to model more accurately the effects of age, which may be non-linearly related to the neurobiological basis of ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Children or adolescents, between 7 and 16 years of age, must have clinical diagnosis of ADHD according to the DSM-5 diagnostic criteria.
* They have to be medication-naïve. They never receive any medication for the treatment of ADHD.
* They and their parents must understand sufficiently to communicate properly with the investigators.
* They must have a Full-Scale Intelligence Quotient(FIQ) score greater than 80.

Exclusion Criteria:

* They have a major psychiatric comorbid disorder, including schizophrenia, schizoaffective disorder, affective disorders, or autism spectrum disorder.
* They have a past history of seizure, or they are taking antiepileptic drugs.
* They have a past history of substance dependence or abuse, including nicotine, alcohol, amphetamine, or any over-the-counter medication.
* They have a past history of major systemic disease.
* They are using Chinese herbs or health supplements.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 120 drug-naïve patients with ADHD, aged 7-16, and 120 age- and sex-matched typically developing controls will be recruited in this project.
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2020-09-19 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
ADHD symptoms | 1 hour
  Subjects will be interviewed by Chinese Version of the Kiddie Epidemiologic version of the Schedule for Affective Disorders and Schizophrenia (K-SADS-E)

SECONDARY OUTCOMES:
Neuropsychological testing | 1.5 hours
  Subjects will be assessed by the Cambridge Neuropsychological Test Automated Battery (CANTAB)
Neuropsychological testing | 15 mins
  Subjects will be assessed by the Continuous Performance Test
Metabolomics profiling | 10 mins
  All the biomarkers are relative ratios. Although all the names of metabolites examined in this study cannot be listed due to the upper limitation of word number (999 characters), the metabolomics profiling includes Hydroxybutyric acid, Undecanedicarboxylic acid, Methyladenosine, Hydroxybutyric acid, Furoylglycine, Hydroxy, Hydroxybutyric acid, Hydroxycaproic acid,Oxoglutarate, Hydroxyisovaleric acid, Hydroxymethylglutaric acid,Indolepropionic acid, Methyladenine, Methylhistidine, Methylindole, Methylxanthine, Pyridylacetic acid, Guanidinobutanoic acid, Dihydrothymine, Aminolevulinic acid, Dodecenoic acid, Hydroxylysine P66-59, Methylcytidine, Acetoacetic acid, Acrylamide, Allose, AMP, Androstenedione, Aspartic acid, Betaine, Bradykinin, Carnitine, Cholic Acid, cis-Aconitate, cis-Fenpropimorph, citric acid, Corticosterone, Creatine, Creatinine, D-Arginine, Decanoylcarnitine, Dehydroascorbic acid, Deoxycholic acid, Deoxyribose, etc.
Brain imaging | 1 hour
  Subjects will be assessed by structural and functional brain imaging, including xoxel-based morphometry, diffusion spectrum imaging, resting-state fMRI, and counting Stroop task fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Study Director — Department of Psychiatry, National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - college of Medicine, National Taiwan University, Taipei